CLINICAL TRIAL: NCT03825367
Title: A Phase I/II Study of Nivolumab in Combination With 5-azacytidine in Pediatric Patients With Relapsed/Refractory Acute Myeloid Leukemia (BMS Reference CA209-9JY)
Brief Title: Nivolumab in Combination With 5-azacytidine in Childhood Relapsed/Refractory AML
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2016-002
Record Dates: First submitted 2019-01-28; First posted 2019-01-31 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: AML, Childhood
Keywords: Relapse; Refractory; Leukemia; Acute; Pediatric; nivolumab; azacytidine
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence; Leukemia | interventions — Nivolumab; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label design (Other): Nivolumab and 5-azacytidine,
  Interventions: Drug: Nivolumab; Drug: 5-azacytidine

INTERVENTIONS:
Drug: Nivolumab — The dose of Nivolumab will be 3 mg/kg which is the adult recommended dose and is the recommended dose in children in the phase 2 portion of COG ADVL1412.
  If 3 mg/kg is not tolerated in combination with 5-azacytidine, the dose will be stepped down to 1 mg/kg.
Drug: 5-azacytidine — 75mg/m2 subcutaneously will be given daily for 7 days on days 1 to 7.

SUMMARY:
This is a phase I/II Study of Nivolumab in Combination with 5-azacytidine in pediatric patients with relapsed/refractory acute myeloid leukemia

DETAILED DESCRIPTION:
This proposed study will be the first to test nivolumab in combination with AZA in pediatric patients with hematologic malignancies. Patients will receive the first dose of nivolumab on day 1 along with AZA. After "chemotherapy priming", a second dose of nivolumab will be given at day 15 which will enhance the effect of nivolumab on the regenerating CD4+ and CD8+ memory T cells.

To establish a recommended Phase II dose (RP2D)of nivolumab in combination with 5-azacytidine in children with relapsed or refractory AML. To assess the clinical activity of Nivolumab in combination with 5-azacytidine in AML patients with M2/M3 disease at study entry.

ELIGIBILITY:
Inclusion Criteria:

Age Patients must be ≥ 1 and ≤30 years of age.

Diagnosis

1. Relapsed or refractory AML with ≥5% blasts (by morphology) in the bone marrow.

   * 1st or greater relapse, OR
   * Failed to go into remission (i.e. refractory) after first or greater relapse, OR
   * Failed to go into remission from original diagnosis after two or more induction attempts.
2. Relapsed or refractory AML with ≤ 5% blasts (by morphology) and MRD positive disease (M1/MRD+): Two serial marrows demonstrating stable or rising MRD ≥ 0.1 % (i.e. not declining). MRD will be determined by multiparameter flow cytometry using AML-associated phenotype markers, or real-time quantitative PCR for AML-associated genetic lesions
3. Patients may have CNS 1 or 2 or other sites of extramedullary disease. No cranial irradiation is allowed during the protocol therapy.
4. Patients with secondary AML are eligible.
5. Patients with DNA fragility syndromes (such as Fanconi anemia, Bloom syndrome) are excluded.
6. Patients with Down Syndrome will be eligible and will be included as an observation cohort

Performance Level Karnofsky > 50% for patients > 16 years of age and Lansky > 50% for patients ≤ 16 years of age.

Prior Therapy Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

A. Myelosuppressive chemotherapy

1. Prior chemotherapy Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. At least 14 days must have elapsed since the completion of the cytotoxic therapy, except Intrathecal chemotherapy.
2. Cytoreduction with hydroxyurea Hydroxyurea can be initiated and continued for up to 24 hours prior to the start of day 1 nivolumab and azacytidine. It is recommended to use hydroxyurea in patients with significant leukocytosis (WBC > 50,000/L) to control blast count before initiation of systemic protocol therapy.

B. Hematopoietic stem cell transplant: Patients who have experienced their relapse after a HSCT are eligible provided they have no evidence of active GVHD, no past history of grade 3 or greater GVHD, and are at least 100 days post-transplant at the time of enrollment. Patients should be off immune suppression for at least 2 weeks (excluding physiologic replacement steroids).

C. Hematopoietic growth factors: It must have been at least 7 days since the completion of therapy with GCSF or other growth factors at the time of enrollment. It must have been at least 14 days since the completion of therapy with pegfilgrastim (Neulasta®).

D. Biologic (anti-neoplastic agent): At least 7 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair

E. Monoclonal antibodies: At least 3 half-lives of the antibody must have elapsed after the last dose of monoclonal antibody. (i.e. Gemtuzumab = 36 days)

F. Immunotherapy: At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines or CAR T-cells.

G. XRT: XRT is prohibited during protocol therapy. No washout period is necessary for radiation given to non-CNS chloromas; ≥ 90 days must have elapsed if prior TBI or craniospinal XRT.

Renal and hepatic function

Patients must have adequate renal and hepatic functions as indicated by the following laboratory values:

A. Adequate renal function defined as: Patient must have a calculated creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73m2 OR a normal serum creatinine based on age/gender in the chart below:

B. Adequate Liver Function Defined as: Direct bilirubin < 1.5 x upper limit of normal (ULN) for age or normal, AND alanine transaminase (ALT) < 5 x ULN for age. The hepatic requirements are waived for patients with known or suspected liver involvement by leukemia. This must be reviewed by and approved by the study chair or vice chair.

Adequate Cardiac Function Defined as: Shortening fraction of ≥ 27% OR ejection fraction of ≥ 50%.

Reproductive Function A. Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed within 24 hours prior to first dose.

B. Female patients with infants must agree not to breastfeed their infants while on this study.

C. Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study and for a minimum of 7 months after study treatment. Women of childbearing potential (WOCBP) receiving nivolumab will be instructed to adhere to contraception for a period of 5 months after the last dose of nivolumab. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of nivolumab.

Informed Consent Patients and/or their parents or legal guardians must be capable of understanding the investigational nature, potential risks and benefits of the study. All patients and/or their parents or legal guardians must sign a written informed consent. Age appropriate assent will be obtained per institutional guidelines. To allow non-English speaking patients to participate in this study, bilingual health services will be provided in the appropriate language when feasible.

Protocol Approval All institutional, FDA, and OHRP requirements for human studies must be met.

Exclusion Criteria:

Patients will be excluded if they have a known allergy or hypersensitivity to nivolumab or AZA used in the study.

Patients will be excluded if they have a systemic fungal, bacterial, viral or other infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment. The patient needs to be off pressors and have negative blood cultures for 48 hours.

Patients will be excluded if there is a plan to administer non-protocol chemotherapy, radiation therapy, or immunotherapy during the study period.

Patients will be excluded if they have significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance with the protocol treatment or procedures, interfere with consent, study participation, follow up, or interpretation of study results.

Patients with DNA fragility syndromes (such as Fanconi anemia, Bloom syndrome) are excluded.

Patients with a known history of severe interstitial lung disease or severe pneumonitis or active pneumonitis that is uncontrolled in the opinion of the treating physician.

Patients who have previously been treated with nivolumab will be excluded.

Patients with a known history of any of the following autoimmune diseases are excluded: (a) patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) (b) patients with a history of rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]).

Patients with organ allografts (such as renal transplant) are excluded.

Patients with known Human Immunodeficiency Virus seropositivity will be excluded.

Known to be positive for hepatitis B by surface antigen expression. Known to have active hepatitis C infection (positive by polymerase chain reaction or on antiviral therapy for hepatitis C within the last 6 months).

Pregnant or breastfeeding.

Acute promyelocytic leukemia (APL).

CNS 3 disease.

Patients who have experienced their relapse after a HSCT and are less than 100 days post-transplant at the time of enrollment, have active GVHD at time of enrollment, have past history of grade 3 or greater GVHD, Patients on immune suppression (excluding physiologic replacement steroids).

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Dose Toxicity | 4 weeks
  Occurrence of dose limiting toxicity (DLT) during Cycle 1 of therapy (Phase I)
Remission | 4 weeks
  Achievement of complete remission (CR/CRp/CRi) at the end of cycle 1

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Columbia University Medical Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Children's Health, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital/Baylor College of Medicine, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No